CLINICAL TRIAL: NCT01903252
Title: A Randomised, Active-Controlled, Double-Blind and Open Label Extensions Study to Evaluate the Efficacy, Long-Term Safety and Tolerability of TP05 3.2g/Day for the Treatment of Active Ulcerative Colitis
Brief Title: TP05 for the Treatment of Mild to Moderate Active Ulcerative Colitis (UC)
Acronym: Precision-UC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tillotts Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TP0503
Record Dates: First submitted 2013-07-09; First posted 2013-07-19 (Estimated); Results first posted 2018-08-08 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Acute Ulcerative Colitis
Keywords: UC
MeSH Terms: interventions — Mesalamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TP05 (Mesalazine) 1600mg (Experimental): week 1 - week 12 (blinded), week 13 - week 38 (OpenLabel)
  Interventions: Drug: TP05
- Asacol 400 mg (Tillotts Pharma) (Active Comparator): week 1 - week 12 (blinded), switch to TP05 for weeks 13-38 (open label)
  Interventions: Drug: Asacol 400 mg

INTERVENTIONS:
Drug: TP05 — 3.2g/day once daily for 12 weeks (blinded), 1.6g/d - 4.8g/d up to week 38 (open label)
  Other Names: Mesalazine 1600 mg
  Arms: TP05 (Mesalazine) 1600mg
Drug: Asacol 400 mg — 3.2g/d twice daily for 12 weeks (blinded), switch to 1.6g/ - 4.8g/d TP05 up to week 38 (open label)
  Other Names: Mesalazine (Tillotts Pharma AG)
  Arms: Asacol 400 mg (Tillotts Pharma)

SUMMARY:
The purpose of this research study was to compare the medication TP05 to the medication Asacol™ for the treatment of ulcerative colitis (UC) and to assess the safety and tolerability of TP05. This study investigated whether TP05 is as good as (non-inferior to) Asacol™(1).

(1)The trademark Asacol™ is registered in over 55 countries as Asacol™ and as Octasa™, Fivasa™, Lixacol™, Asacolon™ in the United Kingdom, France, Spain and Ireland, respectively. The rights to Asacol, including the rights to the trademark, are owned by Tillotts Pharma AG in various countries except for the following: Switzerland, USA, United Kingdom, Canada, Italy, Belgium, the Netherlands and Luxembourg.

DETAILED DESCRIPTION:
This is a Phase 3, randomised, double-blind, active-controlled, multi-centre, non-inferiority trial evaluating the safety and efficacy of 3.2 g of TP05/day compared to 3.2 g/day of Asacol™ with an open label extension to assess the long-term safety and tolerability of TP05 administered over a 26 week period. A total of 817 subjects with mildly to moderately active UC were evaluated. Eligible subjects were randomly assigned in a 1:1 ratio to receive 3.2 g/day of TP05 (administered once daily(OD)) or 3.2 g/day of Asacol™. The primary efficacy outcome was assessed at Week 8. All subjects who respond to TP05/Asacol™ (response or remission) continued receiving blinded study treatment for up to 12 weeks. After that, subjects could enroll in an Open Label Extension (OLE) for 26 weeks duration to receive TP05. Subjects failing to respond to study drug at the Week 8 visit could enroll in the OLE at week 8 and received 4.8 g/day of TP05.

ELIGIBILITY:
Induction phase - Main criteria for inclusion include:

1. Male or non-pregnant, non-lactating females, 18 years of age or older. Females of child bearing potential must have a negative serum pregnancy test prior to randomisation, and must use a hormonal (oral, implantable or injectable) or barrier method of birth control throughout the study. Females unable to bear children must have documentation of such in the source records (i.e., tubal ligation, hysterectomy, or post-menopausal [defined as a minimum of one year since the last menstrual period]).
2. Documented diagnosis of UC with disease extending at least 15 cm from the anal verge.
3. Active UC defined by:

   * a. Mayo score of ≥ 5
   * b. Sigmoidoscopy component score ≥ 2 confirmed by central review and
   * c. Rectal bleeding component score ≥ 1
4. Ability of the subject to participate fully in all aspects of this clinical trial.
5. Written informed consent must be obtained and documented.

Induction Phase - Main criteria for exclusion include:

Subjects who exhibit any of the following conditions are to be excluded from the study:

(1) Severe UC defined by the following criteria: 6 bloody stools daily with one or more of the following:

* a. oral temperature > 37.8 degrees C or > 100.0 degrees F
* b. pulse > 90 beats/min
* c. haemoglobin < 10 g/dL (2) Treatment with oral mesalamine at a dose of > 2.4 g/day within 4 weeks prior to randomisation.

  (3) Treatment with topical therapy (mesalamine or corticosteroids) within 2 weeks prior to randomisation (4) Treatment with systemic or rectal steroids within 4 weeks prior to randomisation.

  (5) Treatment with immunosuppressants within 6 weeks prior to randomisation. (6) Treatment with infliximab or other biologics within 3 months prior to randomisation.

  (7) Treatment with antibiotics within 7 days prior to randomisation. (8) Treatment with probiotics within 7 days prior to randomisation. (9) Treatment with anti-diarrhoeal treatment within 7 days prior to randomisation.

  (10) Treatment with nicotine patch within 7 days prior to randomisation. (11) Received any investigational drug within 30 days prior to randomisation. (12) History of colectomy or partial colectomy. (13) History of definite dysplasia in colonic biopsies. (14) Crohn's disease. (15) Immediate or significant risk of toxic megacolon. (16) Known bleeding disorders. (17) Hypersensitivity to salicylates, aspirin, sulfasalazine or mesalazine. (18) Serum creatinine > 1.5 times the upper limit of the normal range. (19) Aspartate aminotransferase (AST), alanine aminotransferase (ALT), total bilirubin or alkaline phosphatase > 2 times the upper limit of the normal range.

  (20) Serious underlying disease other than UC which in the opinion of the investigator may interfere with the subject's ability to fully participate in the study.

  (21) History of alcohol or drug abuse which in the opinion of the investigator may interfere with the subject's ability to comply with the study procedures.

  (22) Stools positive for Clostridium difficile toxin. (23) Pregnant or lactating women. (24) Prior enrolment in the study.

OLE - Main criteria for inclusion include:

1. Attendance at the Week 8 visit and completion of disease activity assessments prior to enrolment in OLE at Week 12 (responders or remitters) or Week 8 (non-responders).
2. At least 75% compliance with study medication in the induction phase.

OLE - Main criteria for exclusion include:

(1) Withdrawal from the induction phase prior to the Week 8 visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 817 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geert R D'Haens, MD, PhD, Principal Investigator — Alimentiv Inc.
Locations (1):
- Tillotts Pharma AG, Rheinfelden, Baslerstrasse 15, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ma C, Jeyarajah J, Guizzetti L, Parker CE, Singh S, Dulai PS, D'Haens GR, Sandborn WJ, Feagan BG, Jairath V. Modeling Endoscopic Improvement after Induction Treatment With Mesalamine in Patients With Mild-to-Moderate Ulcerative Colitis. Clin Gastroenterol Hepatol. 2022 Feb;20(2):447-454.e1. doi: 10.1016/j.cgh.2020.11.040. Epub 2020 Dec 3. PMID 33279779
- [Derived] Ma C, Sandborn WJ, D'Haens GR, Zou G, Stitt LW, Singh S, Ananthakrishnan AN, Dulai PS, Khanna R, Jairath V, Feagan BG. Discordance Between Patient-Reported Outcomes and Mucosal Inflammation in Patients With Mild to Moderate Ulcerative Colitis. Clin Gastroenterol Hepatol. 2020 Jul;18(8):1760-1768.e1. doi: 10.1016/j.cgh.2019.09.021. Epub 2019 Sep 20. PMID 31546056
- [Derived] D'Haens GR, Sandborn WJ, Zou G, Stitt LW, Rutgeerts PJ, Gilgen D, Jairath V, Hindryckx P, Shackelton LM, Vandervoort MK, Parker CE, Muller C, Pai RK, Levchenko O, Marakhouski Y, Horynski M, Mikhailova E, Kharchenko N, Pimanov S, Feagan BG. Randomised non-inferiority trial: 1600 mg versus 400 mg tablets of mesalazine for the treatment of mild-to-moderate ulcerative colitis. Aliment Pharmacol Ther. 2017 Aug;46(3):292-302. doi: 10.1111/apt.14164. Epub 2017 Jun 1. PMID 28568974

RESULTS

PARTICIPANT FLOW:
Groups:
- TP05 (Mesalazine) 1600 mg: 3.2g/day once daily (OD) for 12 weeks (blinded),
- Asacol (Mesalazine 400 mg): 3.2g/d twice daily for 12 weeks (blinded),
- Extended Induction: Non-responders at week 8 of the induction phase were taken out of the double-blind phase and treated with TP05 4.8g/day OD for another 8 weeks
- 1.6g TP05 (1600 mg) /Day Maintenance Open-Label: Remitters at week 12 of the induction phase received a daily dose of 1.6g OD in the maintenance phase open-label.
- 3.2g TP05 (1600 mg) /Day Maintenance Open-Label: Responders at week 12 of the induction phase remained on a daily dose of 3.2 g OD in the maintenance phase open-label.
- 4.8g TP05 (1600 mg) /Day Maintenance Open-Label: Non-responders at week 12 of the double-blind induction phase as well as non-responders at week 8 of the induction phase who responded after a second 8 weeks of extended induction treatments, were enrolled into the maintenance phase and remained on a daily dose of 4.8g OD.
Period: Double-Blind Induction
Arm/Group | TP05 (Mesalazine) 1600 mg | Asacol (Mesalazine 400 mg) | Extended Induction | 1.6g TP05 (1600 mg) /Day Maintenance Open-Label | 3.2g TP05 (1600 mg) /Day Maintenance Open-Label | 4.8g TP05 (1600 mg) /Day Maintenance Open-Label
Started | 409 | 408 | 0 | 0 | 0 | 0
Completed | 370 | 367 | 0 | 0 | 0 | 0
Not Completed | 39 | 41 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 20 | 18 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 10 | 13 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 3 | 0 | 0 | 0 | 0
Not completed — non-compliance, | 7 | 7 | 0 | 0 | 0 | 0
Period: Extended Induction, Open-Label
Arm/Group | TP05 (Mesalazine) 1600 mg | Asacol (Mesalazine 400 mg) | Extended Induction | 1.6g TP05 (1600 mg) /Day Maintenance Open-Label | 3.2g TP05 (1600 mg) /Day Maintenance Open-Label | 4.8g TP05 (1600 mg) /Day Maintenance Open-Label
Started (This treatment arm was only used in Period 1, double-blind induction phase.) | 0 | 0 (This treatment arm was only used in Period 1, double-blind induction phase.) | 243 (The subjects in this phase were non-responders at week 8 and discontinued the double-blind phase.) | 0 | 0 | 0
Completed | 0 | 0 | 220 | 0 | 0 | 0
Not Completed | 0 | 0 | 23 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 17 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 5 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0
Period: Maintenance, Open-Label
Arm/Group | TP05 (Mesalazine) 1600 mg | Asacol (Mesalazine 400 mg) | Extended Induction | 1.6g TP05 (1600 mg) /Day Maintenance Open-Label | 3.2g TP05 (1600 mg) /Day Maintenance Open-Label | 4.8g TP05 (1600 mg) /Day Maintenance Open-Label
Started (All patients received TP05, three diffrent daily doses: 1.6g, 3.2g, 4.8g) | 0 | 0 | 0 (Period 2 (extended induction) is completed, subjects are newly allocated to Period 3, maintenance.) | 202 (This is period 3, Open-Label Maintenance following on from period 1, the double-blind induction.) | 274 (This is period 3, Open-Label Maintenance following on from period 1, the double-blind induction.) | 199 (This is period 3, Open-Label Maintenance following on from period 1, the double-blind induction.)
Completed | 0 | 0 | 0 | 196 | 253 | 181
Not Completed | 0 | 0 | 0 | 6 | 21 | 18
Not completed — Adverse Event | 0 | 0 | 0 | 3 | 9 | 14
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 6 | 2
Not completed — Other | 0 | 0 | 0 | 2 | 6 | 2

BASELINE CHARACTERISTICS:
Population: Safety Population (SAF)/Intent to Treat (ITT)
Groups:
- TP05 (Mesalazine): 3.2 gram/day (g/d) once daily (OD) for 12 weeks (blinded),
- Asacol (Mesalazine, Tillotts Pharma AG): 3.2g/d twice daily for 12 weeks (blinded),
- Total: Total of all reporting groups
Arm/Group | TP05 (Mesalazine) | Asacol (Mesalazine, Tillotts Pharma AG) | Total
Number analyzed (Participants) | 409 | 408 | 817
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.97 (14.54) | 43.3 (14.11) | 43.5 (14.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 171 | 178 | 349
  Male | 238 | 230 | 468
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 378 | 386 | 764
  Black | 1 | 1 | 2
  Asian or Pacific Islander | 7 | 3 | 10
  Mixed/Other | 0 | 1 | 1
  Not Available | 23 | 17 | 40
Region of Enrollment [Number; unit: participants]
  Belarus | 47 | 49 | 96
  Belgium | 9 | 8 | 17
  Bulgaria | 15 | 15 | 30
  Canada | 15 | 17 | 32
  Czech Republic | 20 | 18 | 38
  Denmark | 20 | 16 | 36
  Finland | 2 | 1 | 3
  Hungary | 17 | 11 | 28
  France | 23 | 16 | 39
  Ireland | 1 | 0 | 1
  Latvia | 22 | 22 | 44
  Lithuania | 26 | 28 | 54
  Norway | 4 | 5 | 9
  Poland | 44 | 48 | 92
  Romania | 2 | 1 | 3
  Russian Federation | 51 | 50 | 101
  Serbia | 18 | 18 | 36
  Slovakia | 2 | 3 | 5
  Spain | 0 | 2 | 2
  Sweden | 1 | 2 | 3
  Ukraine | 59 | 71 | 130
  United Kingdom | 11 | 7 | 18
Mayo Score [Mean (Standard Deviation); unit: units on a scale] — Mayo Score and Partial Mayo Clinic Score (PMCS):
  The Mayo scoring system is a well-established tool for assessing UC disease activity. The Mayo score is the sum of 4 component sub-scores, each ranging from 0 representing no pathology to 3 for severe disease. The 4 component sub-scores are: 1) stool frequency, 2) rectal bleeding, 3) flexible sigmoidoscopy scores, and 4) physician's global assessment. The minimum Mayo Score is 0 (no pathology) and the maximum is 12 (severe disease in all sub-scores).
  units on a scale | 7.7 (1.3) | 7.6 (1.3) | 7.7 (1.3)
Partial Mayo Clinic Score [Mean (Standard Deviation); unit: units on a scale] — Partial Mayo Clinic Score (PMCS) is the sum of the component sub-scores, excluding the endoscopic score. The 3 component sub-scores are: 1) stool frequency, 2) rectal bleeding, and 3) physician's global assessment. The minimum is 0, no pathology and the maximum is 9, severe disease in all sub-scores.
  units on a scale | 5.5 (1.1) | 5.3 (1.1) | 5.4 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Period 1: Clinical and Endoscopic Remission
Description: Mayo Score of <= 2 points with no individual sub-score > 1
Time Frame: Week 8
Population: Per Protocol
Measure: Count of Participants; unit: Participants
Groups:
- TP05 (Mesalazine): 3.2g/day once daily for 12 weeks (blinded),
Arm/Group | TP05 (Mesalazine) | Asacol (Mesalazine, Tillotts Pharma AG)
Number analyzed (Participants) | 388 | 386
Participants | 87 | 95
Statistical Analysis 1: Comparison: TP05 (Mesalazine) vs Asacol (Mesalazine, Tillotts Pharma AG); If the lower limit of the confidence interval was no less than -10% it would be concluded that the test product is non-inferior to the comparator; Test type: Non-Inferiority or Equivalence — Non-inferiority, pre-defined non-inferiority margin 10% A two-sided 95% confidence interval about the difference in proportions was constructed. If the lower limit of the confidence interval was no less than -10% it would be concluded that the test product is non-inferior to the comparator; p = 0.005, Non-inferiority; Risk Difference (RD) = -2.2, 95% CI 2-sided [-8.1 to 3.8]

2. Primary Outcome: Period 2: Clinical Response, Open-Label Extended Induction
Description: A decrease in the PMCS of ≥ 2 points and ≥ 30% from baseline, with a decrease in the rectal bleeding sub-score of ≥ 1 point or absolute rectal bleeding sub-score of 1 or 0.
Time Frame: Week 16
Population: Intent to Treat
Measure: Count of Participants; unit: Participants
Groups:
- Extended Induction: Non-responders to blinded treatment at week 8 of the induction phase (Period 1) were moved to open-label extended induction treatment of an additional 8 weeks (Period 2)
Arm/Group | Extended Induction
Number analyzed (Participants) | 243
Participants | 183
Statistical Analysis 1: Comparison: Extended Induction; Test type: Superiority or Other; Percentag = 75.3, 95% CI 2-sided [69.4 to 80.6]

3. Primary Outcome: Period 3: Clinical Remission
Description: Clinical Remission was defined as a score of 0 points for both stool frequency and rectal bleeding on the Partial Mayo Clinic Score (PMCS)
Time Frame: Week 38
Population: Intent to Treat
Measure: Number; unit: percentage of participant
Groups:
- 1.6g/Day Maintenance Open-Label: Remitters at week 12 of the induction phase (Period 1) received a daily dose of 1.6g in the maintenance open-labe phase ((Period 3)
- 3.2/Day Maintenance Open-Label: Responders at week 12 of the induction phase (Period 1) remaining on a daily dose of 3.2g in the maintenance phase open-label (Period 3)
- 4.8g/Day Maintenance Open-Label: Original non-responders at week 8 of the induction phase (Period 1) who responded to treatment after a second 8 weeks of extended induction open-label (Period 2), were enrolled into the maintenance phase open-label (Period 3) and remained on a daily dose of 4.8g.
Arm/Group | 1.6g/Day Maintenance Open-Label | 3.2/Day Maintenance Open-Label | 4.8g/Day Maintenance Open-Label
Number analyzed (Participants) | 202 | 274 | 199
percentage of participant | 70.3 | 33.9 | 30.7

4. Secondary Outcome: Period 1: Endoscopic Remission
Description: Endoscopic remission was defined as a Mayo endoscopy subscore of 0
Time Frame: Week 8
Population: Per Protocol
Measure: Count of Participants; unit: Participants
Arm/Group | TP05 (Mesalazine) | Asacol (Mesalazine, Tillotts Pharma AG)
Number analyzed (Participants) | 388 | 386
Participants | 36 | 44
Statistical Analysis 1: Comparison: TP05 (Mesalazine) vs Asacol (Mesalazine, Tillotts Pharma AG); Test type: Non-Inferiority or Equivalence — non-inferiority; p < 0.001, Non-inferiority; Risk Difference (RD) = -2.1, 95% CI 2-sided [-6.5 to 2.2]

5. Secondary Outcome: Period 1: Endoscopic Response
Description: Endoscopic response was define as a reduction in the Mayo endoscopic sub score of at least one.
Time Frame: Week 8
Population: Per Protocol
Measure: Count of Participants; unit: Participants
Groups:
- TP05 (Mesalazine): 3.2g/day once daily for 12 weeks (blinded)
- Asacol (Mesalazine, Tillotts Pharma AG): 3.2g/d twice daily for 12 weeks (blinded)
Arm/Group | TP05 (Mesalazine) | Asacol (Mesalazine, Tillotts Pharma AG)
Number analyzed (Participants) | 388 | 386
Participants | 185 | 196
Statistical Analysis 1: Comparison: TP05 (Mesalazine) vs Asacol (Mesalazine, Tillotts Pharma AG); Test type: Non-Inferiority or Equivalence — Non-inferiority; p = 0.026, Non-inferiority; Risk Difference (RD) = -3.1, 95% CI 2-sided [-10.1 to 3.9]

6. Secondary Outcome: Period 1: Clinical Remission
Description: as for outcome 3
Time Frame: Week 8
Population: Per Protocol
Measure: Count of Participants; unit: Participants
Arm/Group | TP05 (Mesalazine) | Asacol (Mesalazine, Tillotts Pharma AG)
Number analyzed (Participants) | 388 | 386
Participants | 92 | 110
Statistical Analysis 1: Comparison: TP05 (Mesalazine) vs Asacol (Mesalazine, Tillotts Pharma AG); Test type: Non-Inferiority or Equivalence — Non-inferiority; p = 0.048, Non-inferiority; Risk Difference (RD) = -4.8, 95% CI 2-sided [-10.9 to 1.4]

7. Secondary Outcome: Period 1: Rectal Bleeding Sub-score of 0
Description: Rectal bleeding sub-score of 0 was defined as a sub score on the rectal bleeding component of the Mayo score
Time Frame: Week 8
Population: Per Protocol
Measure: Count of Participants; unit: Participants
Arm/Group | TP05 (Mesalazine) | Asacol (Mesalazine, Tillotts Pharma AG)
Number analyzed (Participants) | 388 | 386
Participants | 212 | 226
Statistical Analysis 1: Comparison: TP05 (Mesalazine) vs Asacol (Mesalazine, Tillotts Pharma AG); Test type: Non-Inferiority or Equivalence — Non-Inferiority; p = 0.042, Non-inferiortiy; Risk Difference (RD) = -3.9, 95% CI 2-sided [-10.8 to 3.1]

8. Secondary Outcome: Period 1: Clinical and Endoscopic Response
Description: Clinical and Endoscopic Response was defined as a decrease in the Mayo score of ≥3 points from baseline and a reduction of ≥ 30% from baseline with either an accompanying decrease in the rectal bleeding sub-score of at least 1 point or an absolute rectal bleeding sub-score of 0 or 1 at the Week 8 visit. If a subject withdrew from the study prior to Week 8 or their response status was not evaluable due to incomplete and/or invalid data, the subject was considered a non-responder.
Time Frame: Week 8
Population: Per Protocol
Measure: Count of Participants; unit: Participants
Groups:
- TP05 (Mesalazine): 3.2g/day once daily at week 8
- Asacol (Mesalazine): 3.2g/d twice daily at week 8
Arm/Group | TP05 (Mesalazine) | Asacol (Mesalazine)
Number analyzed (Participants) | 388 | 386
Participants | 221 | 236
Statistical Analysis 1: Comparison: TP05 (Mesalazine) vs Asacol (Mesalazine); Test type: Non-Inferiority — Non-Inferiority; p = 0.048, Non-inferiority; Risk Difference (RD) = -4.2, 95% CI 2-sided [-11.0 to 2.7]

9. Secondary Outcome: Period 1: Clinical Remission
Description: as for outcome 3
Time Frame: Week 12
Population: Per Protocol
Measure: Count of Participants; unit: Participants
Arm/Group | TP05 (Mesalazine) | Asacol (Mesalazine, Tillotts Pharma AG)
Number analyzed (Participants) | 388 | 386
Participants | 93 | 113
Statistical Analysis 1: Comparison: TP05 (Mesalazine) vs Asacol (Mesalazine, Tillotts Pharma AG); Test type: Non-Inferiority or Equivalence — Non-inferiority; p = 0.068, Non-inferiority; Risk Difference (RD) = -5.3, 95% CI 2-sided [-11.5 to 0.9]

10. Secondary Outcome: Period 1: Clinical Response
Description: as for outcome 2
Time Frame: Week 12
Population: Per protocol
Measure: Count of Participants; unit: Participants
Arm/Group | TP05 (Mesalazine) | Asacol (Mesalazine, Tillotts Pharma AG)
Number analyzed (Participants) | 388 | 386
Participants | 223 | 233
Statistical Analysis 1: Comparison: TP05 (Mesalazine) vs Asacol (Mesalazine, Tillotts Pharma AG); Test type: Non-Inferiority or Equivalence — Non-inferiority; p = 0.021, Non-inferiortiy; Risk Difference (RD) = -2.9, 95% CI 2-sided [-9.8 to 4.0]

11. Secondary Outcome: Period 1: Rectal Bleeding Score of 0
Description: Rectal bleeding sub-score of 0 was defined as a sub score on the rectal bleeding component of the Mayo score
Time Frame: Week 12
Population: Per Protocol
Measure: Count of Participants; unit: Participants
Arm/Group | TP05 (Mesalazine) | Asacol (Mesalazine, Tillotts Pharma AG)
Number analyzed (Participants) | 388 | 386
Participants | 193 | 205
Statistical Analysis 1: Comparison: TP05 (Mesalazine) vs Asacol (Mesalazine, Tillotts Pharma AG); Test type: Non-Inferiority or Equivalence — Non-inferiority; p = 0.031, Non-inferiortiy; Risk Difference (RD) = -3.4, 95% CI 2-sided [-10.3 to 3.7]

12. Secondary Outcome: Period 1: Clinical Remission at Both Week 8 and 12
Description: as for outcome 3
Time Frame: Week 8 and week 12
Population: Per Protocol
Measure: Count of Participants; unit: Participants
Arm/Group | TP05 (Mesalazine) | Asacol (Mesalazine, Tillotts Pharma AG)
Number analyzed (Participants) | 388 | 386
Participants | 66 | 80
Statistical Analysis 1: Comparison: TP05 (Mesalazine) vs Asacol (Mesalazine, Tillotts Pharma AG); Test type: Non-Inferiority or Equivalence — Non-inferiority; p = 0.013, Non-inferiority; Risk Difference (RD) = -3.7, 95% CI 2-sided [-9.2 to 1.8]

13. Secondary Outcome: Period 1: Clinical Response at Both Week 8 and Week 12
Description: A decrease in the Partial Mayo Score of ≥ 2 points and ≥ 30% from baseline, with a decrease in the rectal bleeding sub-score of ≥ 1 point or absolute rectal bleeding sub-score of 1 or 0.
Time Frame: Week 8 and Week 12
Population: Per Protocol
Measure: Count of Participants; unit: Participants
Arm/Group | TP05 (Mesalazine) | Asacol (Mesalazine, Tillotts Pharma AG)
Number analyzed (Participants) | 388 | 386
Participants | 216 | 230
Statistical Analysis 1: Comparison: TP05 (Mesalazine) vs Asacol (Mesalazine, Tillotts Pharma AG); Test type: Non-Inferiority or Equivalence — Non-inferiority; p = 0.042, Non-inferiority; Risk Difference (RD) = -3.9, 95% CI 2-sided [-10.8 to 3.0]

14. Secondary Outcome: Period 1: Change in Mayo Score From Baseline
Description: Between-Group Difference of Mayo Score, Change from Baseline The changes from baseline to week 8 values in Mayo scores are compared between the two treatment groups.
  The Mayo scoring system is a well-established tool for assessing UC disease activity. The Mayo score is the sum of 4 component sub-scores, each scored on a scale ranging from 0 representing no pathology to 3 for severe disease. The 4 component sub-scores consist of, 1) stool frequency, 2) rectal bleeding, 3) flexible sigmoidoscopy scores, and 4) physician's global assessment. A Mayo score of 0 indicates no pathology and a score of 12, severe disease. Change from Baseline is calculated Baseline-score minus week 8-score. A larger change in Mayo score from baseline when patients experienced acute disease, indicates improvement and treatment success.
Time Frame: Baseline and Week 8
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TP05 (Mesalazine) | Asacol (Mesalazine)
Number analyzed (Participants) | 371 | 375
units on a scale | 3.1 (2.7) | 3.2 (2.6)
Statistical Analysis 1: Comparison: TP05 (Mesalazine) vs Asacol (Mesalazine); Test type: Other; p = 0.557, t-test, 2 sided; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.5 to 0.3]

15. Secondary Outcome: Period 1: Change in Partial Mayo Score From Baseline
Description: Between-Group Difference of Partial Mayo Score, Change from Baseline to Week 8 The Partial Mayo Score is the sum of the component sub-scores, 1) stool frequency, 2) rectal bleeding and 3) physician's global assessment. A partial Mayo Score of 0 indicates no disease and a maximum score of 9 indicates severe symptoms. Change from Baseline is calculated Baseline-score minus week 8-score. A larger change in Partial Mayo Score from Baseline where patients experienced acute disease, indicates improvement and treatment success.
Time Frame: Baseline and Week 8
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TP05 (Mesalazine) | Asacol (Mesalazine)
Number analyzed (Participants) | 387 | 383
units on a scale | 2.5 (2.2) | 2.5 (2.2)
Statistical Analysis 1: Comparison: TP05 (Mesalazine) vs Asacol (Mesalazine); Test type: Other; p = 0.987, t-test, 2 sided; Mean Difference (Net) = 0.00, 95% CI 2-sided [-0.3 to 0.3]

16. Secondary Outcome: Period 1: Change in Stool Frequency Score
Description: Between-Group Difference of Stool Frequency Score, Change from Baseline The changes from baseline to week 8 values in stool frequency will be compared between the two treatment groups. Values for stool frequency range between 0 and 3. A value of 0 indicates normal stool frequency, a value of 3 indicates 5 or more stools than normal. Change from Baseline is calculated Baseline-score minus week 8-score. A large difference between week 8 values and baselines indicates treatment success.
Time Frame: Baseline and Week 8
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TP05 (Mesalazine) | Asacol (Mesalazine)
Number analyzed (Participants) | 387 | 383
units on a scale | 0.9 (1.1) | 0.9 (1.1)
Statistical Analysis 1: Comparison: TP05 (Mesalazine) vs Asacol (Mesalazine); Test type: Other; p = 0.455, t-test, 2 sided; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.1 to 0.2] — The result of the mean difference is not corresponding to the values in the table due to rounding as specified in the Statistical Analysis Plan (SAP)

17. Secondary Outcome: Period 1: Change in Rectal Bleeding Score From Baseline
Description: Between-Group Difference of Rectal Bleeding Score, Change from Baseline The changes from baseline to week 8 values in rectal bleeding scores will be compared between the two treatment groups. A value of 0 indicates no rectal bleeding, a value of 3 indicates only blood is passing. Change from Baseline is calculated Baseline-score minus week 8-score. A large difference at week 8 compared to baseline is indicative of treatment success.
Time Frame: Baseline and Week 8
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TP05 (Mesalazine) | Asacol (Mesalazine)
Number analyzed (Participants) | 387 | 383
units on a scale | 0.9 (0.8) | 1.0 (0.8)
Statistical Analysis 1: Comparison: TP05 (Mesalazine) vs Asacol (Mesalazine); Test type: Other; p = 0.937, t-test, 2 sided; Mean Difference (Net) = -0.00, 95% CI 2-sided [-0.1 to 0.1] — The apparent difference between the values in the table and the mean difference is due to rounding as defined in the SAP

18. Secondary Outcome: Period 1: Change in Physician Global Assessment Score From Baseline
Description: Between-Group Difference of Physician Global Assessment Score, Change from Baseline.
  The changes from baseline to week 8 values in the Physician Global Assessment score will be compared between the two treatment groups. A value of 0 means no pathology and a value of 3 means severe disease. Change from Baseline is calculated Baseline-score minus week 8-score. A large difference between baseline to week 8 indicates treatment success.
Time Frame: Baseline and Week 8
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TP05 (Mesalazine) | Asacol (Mesalazine)
Number analyzed (Participants) | 387 | 383
units on a scale | 0.6 (0.8) | 0.7 (0.8)
Statistical Analysis 1: Comparison: TP05 (Mesalazine) vs Asacol (Mesalazine); Test type: Other; p = 0.357, t-test, 2 sided; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.2 to 0.1]

19. Secondary Outcome: Period 1: Change in Endoscopic Score From Baseline
Description: Between-Group Difference of Endoscopic Score, Change from Baseline. The changes from baseline to week 8 values in sigmoidoscopic (mucosal) appearance scores will be compared between the two treatment groups. A value of 0 in the endoscopic score means normal or inactive disease and a value of 3 means severe disease. Change from Baseline is calculated Baseline-score minus week 8-score. A large difference between baseline to week 8 indicates treatment success.
Time Frame: Baseline and Week 8
Population: Per Protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TP05 (Mesalazine) | Asacol (Mesalazine)
Number analyzed (Participants) | 371 | 375
units on a scale | 0.5 (0.9) | 0.6 (0.8)
Statistical Analysis 1: Comparison: TP05 (Mesalazine) vs Asacol (Mesalazine); Test type: Other; p = 0.099, t-test, 2 sided; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.2 to 0.0]

20. Secondary Outcome: Period 2: Clinical Remission
Description: as for outcome 3
Time Frame: Week 16
Population: Intent to Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Extended Induction
Number analyzed (Participants) | 243
Participants | 53
Statistical Analysis 1: Comparison: Extended Induction; Test type: Other; Percentage = 21.8, 95% CI 2-sided [16.8 to 27.5]

21. Secondary Outcome: Period 2: Rectal Bleeding Sub-score of 0
Description: Percentage of patients achieving the endpoint rectal bleeding sub-score of 0
Time Frame: Week 16
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Extended Induction
Number analyzed (Participants) | 243
Participants | 146
Statistical Analysis 1: Comparison: Extended Induction; Test type: Other; Percentage = 60.1, 95% CI 2-sided [53.6 to 66.3]

22. Secondary Outcome: Period 2: Stool Frequency 0
Description: Percentage of patients achieving the endpoint stool frequency sub-score of 0
Time Frame: Week 16
Population: Intent to Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Extended Induction
Number analyzed (Participants) | 243
Participants | 64
Statistical Analysis 1: Comparison: Extended Induction; Test type: Other; Percentage = 26.3, 95% CI 2-sided [20.9 to 32.3]

23. Secondary Outcome: Period 2: Urgency
Description: Percentage of patients achieving an Urgency Score of 0. A score of 0 indicates no urgency reported in any of the three days prior to the visit at week 16. A score of 1 indicates urgency reported in any of the three days prior to the visits.
Time Frame: Week 16
Population: Indent to Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Extended Induction
Number analyzed (Participants) | 243
Participants | 109
Statistical Analysis 1: Comparison: Extended Induction; Test type: Other; Percentage = 44.9, 95% CI 2-sided [38.5 to 51.3]

24. Secondary Outcome: Period 2: UC-Related Complications
Description: Percentage of Patients Experiencing Complications related to UC
Time Frame: Week 16
Population: Intent to Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Extended Induction
Number analyzed (Participants) | 243
Participants | 0.0
Statistical Analysis 1: Comparison: Extended Induction; Test type: Other; Percentage = 0.00, 95% CI 2-sided [0.0 to 1.5]

25. Secondary Outcome: Period 3: Clinical Response
Description: as for outcome 2
Time Frame: Week 38
Population: Intent to Treat
Measure: Number; unit: percentage of participants
Arm/Group | 1.6g/Day Maintenance Open-Label | 3.2/Day Maintenance Open-Label | 4.8g/Day Maintenance Open-Label
Number analyzed (Participants) | 202 | 274 | 199
percentage of participants | 94.1 | 83.9 | 78.4

26. Secondary Outcome: Period 3: Clinical and Endoscopic Remission
Description: Mayo Score of <= 2 points with no individual sub-score > 1
Time Frame: Week 38
Population: Intent to Treat
Measure: Number; unit: percentage of participants
Arm/Group | 1.6g/Day Maintenance Open-Label | 3.2/Day Maintenance Open-Label | 4.8g/Day Maintenance Open-Label
Number analyzed (Participants) | 202 | 274 | 199
percentage of participants | 65.8 | 39.4 | 29.6

27. Secondary Outcome: Period 3: Clinical and Endoscopic Response
Description: Both has to be achieved, Clinical and Endoscopic Response which is defined by a decrease from baseline in the Mayo score of ≥ 3 points and > 30% of the baseline score, with an accompanying decrease in the rectal bleeding sub-score of ≥ 1 point or an absolute rectal bleeding sub-score of 0 or 1.
Time Frame: Week 38
Population: Intent to Treat
Measure: Number; unit: percentage of participants
Arm/Group | 1.6g/Day Maintenance Open-Label | 3.2/Day Maintenance Open-Label | 4.8g/Day Maintenance Open-Label
Number analyzed (Participants) | 202 | 274 | 199
percentage of participants | 89.6 | 78.1 | 69.3

28. Secondary Outcome: Period 3: Endoscopic Remission
Description: Percentage of each dose group achieving an endoscopy sub score of 0
Time Frame: Week 38
Population: Intent to Treat
Measure: Number; unit: percentage of participants
Arm/Group | 1.6g/Day Maintenance Open-Label | 3.2/Day Maintenance Open-Label | 4.8g/Day Maintenance Open-Label
Number analyzed (Participants) | 202 | 274 | 199
percentage of participants | 37.6 | 32.4 | 13.6

29. Secondary Outcome: Period 3: Endoscopic Response
Description: Endoscopic response was define as a reduction in the Mayo endoscopic sub score of at least one.
Time Frame: Week 38
Population: Intent to Treat
Measure: Number; unit: percentage of participants
Arm/Group | 1.6g/Day Maintenance Open-Label | 3.2/Day Maintenance Open-Label | 4.8g/Day Maintenance Open-Label
Number analyzed (Participants) | 202 | 274 | 199
percentage of participants | 73.8 | 58.8 | 53.3

30. Secondary Outcome: Period 3: Rectal Bleeding Sub Score of 0
Description: Percentage of each dose group achieving the endpoint rectal bleeding subscore 0
Time Frame: Week 38
Population: Intent to Treat
Measure: Number; unit: percentage of participants
Arm/Group | 1.6g/Day Maintenance Open-Label | 3.2/Day Maintenance Open-Label | 4.8g/Day Maintenance Open-Label
Number analyzed (Participants) | 202 | 274 | 199
percentage of participants | 88.1 | 76.3 | 74.9

31. Secondary Outcome: Period 3: Stool Frequency Sub-score 0
Description: Patients achieving a Stool Frequency sub-score of 0
Time Frame: Week 38
Population: Intent to Treat
Measure: Count of Participants; unit: Participants
Arm/Group | 1.6g/Day Maintenance Open-Label | 3.2/Day Maintenance Open-Label | 4.8g/Day Maintenance Open-Label
Number analyzed (Participants) | 202 | 274 | 199
Participants | 148 | 101 | 66

32. Secondary Outcome: Period 3: No Urgency
Description: No urgency is a score of 0 and indicates that patients did not report urgency during any of the three days prior to the visit at week 38. A score of 1 indicates that urgency was reported during any of these three days.
Time Frame: Week 38
Population: Intent to Treat
Measure: Count of Participants; unit: Participants
Arm/Group | 1.6g/Day Maintenance Open-Label | 3.2/Day Maintenance Open-Label | 4.8g/Day Maintenance Open-Label
Number analyzed (Participants) | 202 | 274 | 199
Participants | 161 | 173 | 109

33. Secondary Outcome: Period 3: UC-Related Complications
Description: Percentage of Patients with Complications related to UC
Time Frame: Week 38
Population: Intent to Treat
Measure: Count of Participants; unit: Participants
Groups:
- 1.6g/Day Maintenance Open-Label: Remitters at week 12 of the induction phase (Period 1) received a daily dose of 1.6g in the maintenance open-labe phase (Period 3)
Arm/Group | 1.6g/Day Maintenance Open-Label | 3.2/Day Maintenance Open-Label | 4.8g/Day Maintenance Open-Label
Number analyzed (Participants) | 202 | 274 | 199
Participants | 3 | 2 | 1

ADVERSE EVENTS:
Time Frame: 2 years, 11 months
Description: Adverse Events (AEs) were analysed for each arm of the double-blind Induction Phase, for the Open-Label Extended Induction Phase and combined for the double-blind Induction Phase and the Open-Label Maintenance Phase but not for the Open-Label Maintenance Phase separately. In adding safety results of the Maintenance Phase to the safety results of the Induction Phase ensured that one occurence of an AE was counted as one AE and not as two when AEs continued from one phase to the other.
Groups:
- TP05/TP05: Double-blind Induction Phase: TP05, and Open-Label Maintenance Phase: TP05
- Asacol/TP05: Double-blind Induction Phase: Asacol, and Open-Label Maintenance Phase: TP05
- TP05 Extended Induction: Extended Induction only, Open-Label
- TP05; Asacol: Double-blind Induction Phase only
Arm/Group | TP05/TP05 | Asacol/TP05 | TP05 Extended Induction | TP05 | Asacol
Serious Adverse Events (participants affected / at risk) | 24/409 | 18/408 | 3/243 | 9/409 | 7/408
Other Adverse Events (participants affected / at risk) | 58/409 | 75/408 | 0/243 | 26/409 | 22/408
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TP05/TP05 (N=409) | Asacol/TP05 (N=408) | TP05 Extended Induction (N=243) | TP05 (N=409) | Asacol (N=408)
Deterioration ulcerative colities (Gastrointestinal disorders) | 9 (10) | 6 (7) | 0 (0) | 4 (5) | 4 (4)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1) — Iron deficiency
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium dificile (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertensive heart disease (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Artrial fibrilation (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic tonsilitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cryoglobulinemic vasculitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flue (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Chronic pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Unstable angina (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herniated disc (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Perichondritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Acute heamorrhagic cystitis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal septum deformation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diabetes melitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fading fetus (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TP05/TP05 (N=409) | Asacol/TP05 (N=408) | TP05 Extended Induction (N=243) | TP05 (N=409) | Asacol (N=408)
Worsening of UC (Gastrointestinal disorders) | 58 (59) | 75 (75) | 0 (0) | 26 (27) | 22 (22) — Symptoms of active ulcerative colitis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No